CLINICAL TRIAL: NCT03323697
Title: The Chinese Herb SZ-05 for the Treatment of Depression and Anxiety Disorders; Efficiency, Safety and Biological Correlates
Brief Title: Chinese Herb for the Treatment of Depression and Anxiety Disorders
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mazra Mental Health Center (Other)
Collaborators: The Academic College of Tel-Aviv Yaffo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MZR-0018-016
Record Dates: First submitted 2017-10-01; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Depression, Anxiety
Keywords: Depression; Anxiety; Herbal Medicine; Chinese Medicine; Hamilton Scale; SSRI
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herbal (Experimental): SZ-05 (2.5 gr; 3 capsules twice a day)
  Interventions: Other: SZ-05
- Selective serotonin reuptake inhibitor (Active Comparator): Escitalopram (10 mg capsule plus 5 placebo capsules)
  Interventions: Drug: Escitalopram Pill

INTERVENTIONS:
Other: SZ-05 — 2.5g a day (3 capsules twice a day)
  Other Names: no other names
  Arms: Herbal
Drug: Escitalopram Pill — 10 mg capsule plus 5 placebo capsules
  Other Names: no other names
  Arms: Selective serotonin reuptake inhibitor

SUMMARY:
Anxiety and depression are currently among the ten most important public health concerns, and in recent years, have reached epidemic proportions. Anxiety is recognized as the main risk factor for many diseases including cardiovascular, metabolic and neuropsychiatric disorders. Current anxiolytic medications have a relatively low success rate (~50%) and are associated with many deleterious side-effects. The investigators aim to investigate the efficacy, safety, and tolerability of a novel herbal treatment on anxiety and depression symptoms in a 6-week double-blind randomized trial.

DETAILED DESCRIPTION:
The relationship between depression and anxiety disorders has long been described, and comorbid depression and anxiety are highly prevalent conditions. The current study will focus on mild to moderate depressive and anxiety symptoms and include a variety of individuals from the depression and anxiety spectrum disorders.The objectives of the current study are to evaluate the antidepressant and anxiolytic efficacy of SZ-05 treatment in a 6-week double-blind randomized trial, and underlying the molecular mechanisms.

Clinical trial study design:

A randomized, double-blind controlled trial will be performed. Patients will be randomized to SZ-05 (2.5 gr (14); 2-3 capsules twice a day, and 1 placebo capsule) or escitalopram (10 mg capsule plus 5 placebo capsules at the same regime as SZ-05) daily treatment at a ratio of 2:1. Overall the study will be conducted for 8 weeks, and will include six weeks of double-blind controlled trial, followed by two weeks of escitalopram treatment. 30 patients will be enrolled to each arm of the trial (overall 60 patients will be recruited). After baseline evaluation and signing informed consent, subjects will be asked to fill a socio-demographic questionnaire, and to undergo a clinical differential diagnosis using the Symptoms Check List (SCL)-90, Clinical Global Impression (CGI), Hamilton anxiety rating scale (HAM-A), Hamilton depression rating scale (HAM-D), Sheehan Disability Scale (SDS), and two visual analogue scales (VAS)- general anxiety, and mood. Subjects will be monitored at baseline and every two weeks for six weeks, and every week in the last two weeks of the trial using HAM-A, HAM-D, VASs and SDS. Adverse effects will be documented every evaluation using the Treatment Emergent Symptom Scale. Subjects will be monitoring for heart rate and blood pressure at baseline and every week till the end of the trial. The herbal treatment and escitalopram will be added to the current drug treatment (non-antidepressant). Any change in the patient non-antidepressant treatment is required to be reported to the study personnel.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes suffering from mild to moderate depressive episode of major depressive disorder (MDD) according to Diagnostic and Statistical Manual Diploma in Social Medicine (DSM)-V.
* Subjects of both sexes meeting the DSM-V criteria for dysthymia.
* Patients of both sexes meeting the DSM-V criteria for Generalized Anxiety Disorder (GAD), Panic Disorder and Social Anxiety Disorder, Adjustment disorder.
* Age 18-65.
* Not receiving antidepressant drugs.
* Hamilton Depression Rating Scale (HAM-D) scores are ≥8 and ≤ 18.
* Hamilton Anxiety Rating Scale (HAM-A) scores ≥17 and ≤ 30.

Exclusion Criteria:

* Current active and persistent substance and/or alcohol abuse.
* Mental retardation
* Other major psychiatric disorders: Psychosis, Severe MDD and Bipolar disorder
* Suicide ideation
* Pregnancy
* Systolic Blood Pressure < 100 mm Hg
* Heart rate < 60 times/min
* Patient with medical history of cardiac palpitation and other cardiac diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety symptoms | Subjects will be monitored at baseline and every two weeks for six weeks
  Changes in HAM-A rates
Depressive symptoms | Subjects will be monitored at baseline and every two weeks for six weeks
  Changes in HAM-D rates

SECONDARY OUTCOMES:
Wellbeing | Subjects will be monitored at baseline and every two weeks for six weeks
  Changes in SDS rate

CONTACTS AND LOCATIONS:
Overall Officials: Efrat City, MD, Principal Investigator — Mazor MHC
Locations (1):
- Mazor MHC, Acre, Israel

IPD SHARING:
Plan to Share IPD: No